CLINICAL TRIAL: NCT03938922
Title: A Multicenter, Open Label Study to Evaluate Tolerability and Efficacy of Orally Administered ENT-01 for the Treatment of Parkinson's Disease Dementia.
Brief Title: A Study to Evaluate ENT-01 for the Treatment of Parkinson's Disease Dementia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Compound will not be studied for indication
Sponsor: Enterin Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENT-01-1b-19-01
Record Dates: First submitted 2019-04-18; First posted 2019-05-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Dementia
Keywords: PDD; parkinson's disease-related dementia
MeSH Terms: conditions — Parkinson Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Treatment (Experimental): ENT-01 tablet will be taken once daily by mouth.
  Interventions: Drug: Active Investigational Treatment ENT-01

INTERVENTIONS:
Drug: Active Investigational Treatment ENT-01 — ENT-01 will be administered in tablet form, once daily.
  Other Names:
  ENT-01

SUMMARY:
This study will be conducted as a multi-center, open label study in the US. There will be 40 patient to receive the active investigational product.

DETAILED DESCRIPTION:
The study will be conducted on an out-patient basis. Each patient will have 5 visits to the clinic: a screening visit, a randomization visit, 1 followup visit, 1 end of treatment visit, and 1 end of study visit.

Patients will be allowed to adjust their dosing, based upon protocol specifications. Rescue medications will be provided to all patients to ensure they move their bowels on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-90 years, both genders
* Patients or care-giver must provide informed consent and be willing and able to comply with study procedures.
* Patients must be diagnosed with Parkinson's disease defined as the presence of at least three of the following cardinal features, in the absence of alternative explanations or atypical features: rest tremor, rigidity, bradykinesia and/or akinesia, postural and gait abnormalities.
* Patients must have dementia as defined by (1) decline in cognitive function and (2) functional impairment, which together in, in the opinion of the investigator, has resulted in a clinical diagnosis of dementia.
* MoCA < 24 in support of a dementia diagnosis
* Have a reliable and actively involved caregiver who must be able to communicate in English and be willing to comply with protocol requirements.
* If on anti-parkinsonian agents, participants must be on stable dosage for at least 4 weeks prior to baseline.
* If on medications enhancing cognition (rivastigmine, galantamine, donepezil, memantine), participants must be on stable dosage for at least 8 weeks prior to baseline.
* If on antidepressant medications, participants must be on stable dosage for at least 4 weeks prior to baseline.
* If on clozapine, pimavanserin or quetiapine to address drug-induced or disease-related psychosis, participants must be on stable dosage for 4 weeks prior to baseline.
* Female patients of childbearing potential must have negative serum or urine pregnancy tests and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. A vasectomized partner will be allowed as one in conjunction with another single-barrier method.
* Female patients unable to bear children must have this documented in the case report form (CRF) (i.e., tubal ligation, hysterectomy, or postmenopausal [defined as a minimum of one year since the last menstrual period]). Post-menopausal status will be confirmed by follicle stimulating hormone (FSH) in women less than 60 years of age.

Exclusion Criteria:

* Patient or caregiver unable or unwilling to provide informed consent or to comply with study procedures.
* Unable to withdraw proton pump inhibitors at the end of run-in period.
* Unable to withdraw from anti-cholinergics at the beginning of the run-in period
* Any clinically significant abnormalities on screening laboratories or physical examination requiring further evaluation or treatment.
* Neurological disorder other than Parkinson's disease that in the opinion of the investigator might interfere with the conduct of the study
* Females who are pregnant or breastfeeding
* History of excessive alcohol use or substance abuse
* Psychotic disorder was present before the diagnosis of Parkinson's disease
* Patient or caregiver unable to administer daily oral dosing of study drug
* Caregiver unwilling or unable to unable to complete stool diary, dispense study medication and accompany the patient to all visits
* Participation in an investigational drug trial within the month prior to dosing in the present study.
* A compromised gastrointestinal system which includes: Structural, metabolic, or functional GI diseases or disorders; History of major GI surgery within 30 days (a history of cholecystectomy, polypectomy, hernia repair, appendicectomy, gastric surgery for peptic ulcer and gastric banding for obesity are not exclusionary as long as they were performed more than 30 days before the screening visit. Partial or complete colectomy is exclusionary).
* Review of Screening period diaries indicates either of the following: Fewer than 11 days of diary completion; More than 5 complete spontaneous bowel movements per week based upon the average Complete Spontaneous Bowel Movement (CSBM) rate reported during the Screening Period.
* Any other reason, which in the opinion of the investigator would confound proper interpretation of the study.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Cognition Improvement by Dementia Severity Rating Scale (DSRS) - Primary Outcome | 10 weeks
  To determine the safety and efficacy of repeated oral doses of ENT-01 in improving cognition in patients with Parkinson's disease dementia, measured by the Dementia Severity Rating Scale (DSRS).
  The DSRS Test is used to track changes in cognitive status over time. Its five subscales provide additional information on specific abilities: Attention, Initiation/Perseveration, Construction, Conceptualization, and Memory.
  The score ranges from 0 to 54, with 0-18 being mild, 19-36 being moderate and 37-54 being severe. Improvements would be indicated by lower scores from baseline to end of fixed dose period.

SECONDARY OUTCOMES:
Change from Baseline in Montreal Cognitive Assessment (MOCA) - Secondary Outcomes | 10 weeks
  To determine the effect of repeated oral doses of ENT-01 in improving cognition in patients with Parkinson's disease Dementia, measured by an improvement in the Montreal Cognitive Assessment (MOCA) from baseline.
Change from Baseline to the End of the Fixed Dose Period in Symptoms Adapted for Parkinson's Disease (SAPS-PD) - Secondary Outcomes | 10 weeks
  To determine the effect of repeated oral doses of ENT-01 in improving the frequency and/or severity of hallucinations/delusions during the Fixed Dose period over baseline in patients with Parkinson's disease Dementia.
  Improvement is defined as 2.33 points or greater reduction in score from baseline on the SAPS-PD.
Change from Baseline to the End of the Fixed Dose Period in Neuropsychiatric Inventory (NPI) and Caregiver Distress (NPI-D) - Secondary Outcomes | 10 weeks
  To determine the effect of repeated oral doses of ENT-01 in patients with Parkinson's disease Dementia, measured by an improvement in total score for behavioral impairment from baseline to the end of fixed dose for the NPI and NPI-D.
  The NPI total score is calculated by adding the scores of the domains (each domain scores ranges from 0 to 144, with higher scores indicating greater behavioral impairment.
  The caregiver distress scores in each of the domains are not included in the NPI total score. The caregiver distress (NPI-D) total score is calculated by adding scores of caregiver distress in each of the domains (score ranges from 0 to 5 in each domain). The NPID total score ranges from 0 to 60 with higher scores indicating greater distress.
Change from Baseline to the End of the Fixed Dose Period in Parkinson's Disease Questionnaire-39 (PDQ-39) - Secondary Outcomes | 10 weeks
  To determine the effect of repeated oral doses of ENT-01 in patients with Parkinson's disease Dementia, measured by an improvement in behavioral impairment, cognition, and social function by having lower scores for the PDQ-39 from baseline to the end of fixed dose.
  The PDQ-39 assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. Lower scores indicate better quality of life. There is a 5-point ordinal system for scoring - 0 is never, and 4 is always.

OTHER OUTCOMES:
To compare the effect of ENT-01 on motor and non-motor symptoms of Parkinson's disease including Movement Disorder Society - Unified Parkinsons' Disease Rating Scale (MDS-UPDRS). | 10 weeks
  The additional efficacy endpoints of the study are the change from baseline in each of the following tests during the Fixed Dose Period (FDP). Baseline is defined as the end of the screening period (Visit 2). Improvement is indicated by lower total scores for the MDS-UPDRS.
  The standard four-part MDS-UPDRS will be administered to determine whether there is any improvement in scores during the treatment period. Motor deterioration will be assessed from Part 3 of the MDS-UPDRS, but total score will also be reported (sum of Parts 1, 2, and 3).
To compare the effect of ENT-01 on non-motor symptoms of Parkinson's disease for skin-temperature determined Circadian rhythm and weight. | 10 weeks
  The additional efficacy endpoints of the study are the changes in skin temperature using an I-button attached to a wrist band. The I-button will be worn throughout the study, from Visit 1 to Visit 5.
To compare the effect of ENT-01 on non-motor symptoms of Parkinson's disease for weight. | 10 weeks
  Body weight will be measured from Visit 1 to Visit 5.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zasloff, MD, Ph.D, Study Chair — Enterin Inc.; Denise Barbut, MD, FRCP, Study Chair — Enterin Inc.
Locations (3):
- United States (3):
  - Neuro Pain Medical Center, Fresno, California
  - Evolution Research Group - Neuroscience Research Institution, Toms River, New Jersey
  - Elias Research - Neurology Diagnostics Research, Dayton, Ohio